CLINICAL TRIAL: NCT00559676
Title: Phase 4 Study to Characterize and Evaluate Markers of Chemoresistance in Patients With Metastatic Colorectal Cancer
Brief Title: Study of Biomarkers in Patients Undergoing Chemotherapy for Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospital Regional Universitaire de Limoges (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: CDR0000574159; CHUL-BIO-COLON; INCA-RECF0356
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2009-07

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Fluorouracil; Irinotecan; Leucovorin; Oxaliplatin

INTERVENTIONS:
Drug: capecitabine
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium
Drug: oxaliplatin
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Studying samples of blood and tumor tissue in the laboratory from patients with cancer receiving chemotherapy may help doctors understand the effect of chemotherapy on biomarkers. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This phase IV trial is studying biomarkers in patients undergoing chemotherapy for metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Research the oncogenetic parameters and pharmacogenetic and pharmacokinetic predictors of therapeutic response and toxic effects.

Secondary

* Study the correlations between the pharmacogenetic and pharmacokinetic parameters.
* Study the predictive value of these parameters on disease-free and overall survival.

OUTLINE: This is a multicenter study.

Patients receive 1 of 4 chemotherapy regimens:

* Regimen 1: Fluorouracil and leucovorin calcium
* Regimen 2: Capecitabine and leucovorin calcium
* Regimen 3: Irinotecan hydrochloride
* Regimen 4: Oxaliplatin Tumor and blood samples are collected before the start of chemotherapy and are examined by pharmacogenetic analysis. Clinical and biological parameters are also studied. Blood samples are also collected during the first course of chemotherapy for pharmacokinetic studies.

After completion of study therapy, patients are followed periodically for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic colorectal cancer

  * Unresectable metastatic disease must be confirmed histologically if > 2 years since primary diagnosis
* Measurable metastatic disease > 1 cm by spiral CT scan or > 2 cm by other methods
* Scheduled to receive first-line chemotherapy for metastatic disease

  * Chemotherapy must include fluorouracil, capecitabine, irinotecan hydrochloride, or oxaliplatin
* No inadequate or unusable tissue as the only tissue available
* No known brain metastases or meningeal disease

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* No contraindication to chemotherapy
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other severe pathology that is likely to worsen during therapy
* No dementia or severely impaired mental condition
* No geographical or psychological reasons that would preclude treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior therapy for metastatic cancer
* Prior adjuvant chemotherapy allowed
* Concurrent bevacizumab or other monoclonal antibody therapy allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2005-03; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Oncogenetic parameters
Pharmacogenetic and pharmacokinetic predictors of therapeutic response and toxic effects

SECONDARY OUTCOMES:
Correlations between the pharmacogenetic and pharmacokinetic parameters
Predictive value of pharmacogenetic and pharmacokinetic parameters on disease-free and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Tubiana-Mathieu, MD, Study Chair — Centre Hospital Regional Universitaire de Limoges
Locations (1):
- Centre Hospital Regional Universitaire de Limoges, Limoges, France

REFERENCES:
- [Derived] Deyme L, Barbolosi D, Mbatchi LC, Tubiana-Mathieu N, Ychou M, Evrard A, Gattacceca F. Population pharmacokinetic model of irinotecan and its four main metabolites in patients treated with FOLFIRI or FOLFIRINOX regimen. Cancer Chemother Pharmacol. 2021 Aug;88(2):247-258. doi: 10.1007/s00280-021-04255-9. Epub 2021 Apr 28. PMID 33912999